CLINICAL TRIAL: NCT05537155
Title: Buccal Acupuncture for Delirium Treatment in Older Patients Recovering From Orthopedic Surgery: a Randomized Controlled Trial
Brief Title: Buccal Acupuncture for Delirium Treatment in Older Patients Recovering From Orthopedic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We do not have enough physicians who are authorized to perform buccal acupuncture in both hospitals.
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-220
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Older Patients; Orthopedic Surgery; Postoperative Delirium; Acupuncture; Treatment
Keywords: Older patients; Orthopedic surgery; Postoperative delirium; Buccal acupuncture; Treatment effects
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buccal acupuncture (Experimental): Buccal acupuncture will be performed in addition to routine care.
  Interventions: Procedure: Buccal acupuncture in addition to routine care
- Routine care (Active Comparator): Routine care will be provided.
  Interventions: Other: Routine care

INTERVENTIONS:
Procedure: Buccal acupuncture in addition to routine care — Acupuncture will be performed at a depth of 10 mm, with the needle retaining for 20 min, in addition to routine care. Bilateral acupoints include "Tou", "Shangjing", "Jing", "Bei", and "Sanjiao". Unilateral acupoints is related to surgical sites and include "Kuan" in hip joint replacement surgery and "Xi" in knee joint replacement surgery. Patients with agitation will be treated first until agitation is controlled before acupuncture is performed.
  Arms: Buccal acupuncture
Other: Routine care — Routing care includes the following: (1) remove the precipitating cause and treat the primary disease; and (2) supportive care, including reorientation and cognitive stimulation, sleep enhancement, early mobility and exercise, vision and hearing optimization, family engagement and empowerment, and early oral intake and nutrition.
  Arms: Routine care

SUMMARY:
This study is designed to test the hypothesis that, for older orthopedic patients who developed postoperative delirium, combining buccal acupuncture with routine care will shorten delirium duration and relieve delirium severity.

DETAILED DESCRIPTION:
Delirium is an acute, transient central nervous system dysfunction characterized by fluctuating disturbances of attention, consciousness, and cognitive function. Delirium is common in older patients following surgery. The incidence of postoperative delirium ranges from 12.0% to 23.8% in older patients; the incidence of delirium is about 10.7-17.6% in older patients after joint replacement surgery. The occurrence of delirium is associated with worse outcomes, including increased early postoperative complications, prolonged hospital-stay, and increased in-hospital mortality, as well as long-term decline in cognitive function, quality of life, and survival duration.

Clinical use of acupuncture has a long history in China. Buccal acupuncture therapy is a microneedle technique and provides treatment for systemic diseases by acupuncturing specific acupoints in the cheek. Acupuncture is also used for delirium treatment. Studies of older patients who developed delirium in internal medicine wards found that, compared with routine care alone, combining routine care with acupuncture relieved delirious symptoms and severity more efficaciously. However, evidence in this aspect is limited. We suppose that, for older orthopedic patients who developed postoperative delirium, combining buccal acupuncture with routine care will shorten delirium duration and relieve delirium severity.

ELIGIBILITY:
Inclusion criteria:

* Aged ≥65 years, but <90 years.
* After knee or hip replacement surgery.
* Diagnosed with delirium in the morning of enrollment.

Exclusion criteria:

* Refuse to participate in the study.
* Presence of any contraindications to acupuncture, such as puncture site infections or platelet count ≤20×10^9/L.
* Preoperative history of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis.
* Inability to communicate due to coma, profound dementia, or language barrier, or inability to cooperate with treatment due to agitation.
* American Society of Anesthesiologists physical status grade ≥V, or estimated survival ≤24 h.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Number of delirium-free days within 5 days | Up to 5 days after enrollment
  Delirium will be assessed twice daily (8:00-10:00 am, 18:00-20:00 pm) with the 3D-Confusion Assessment Method (3D-CAM) for non-intubated patients or the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) for intubated patients.

SECONDARY OUTCOMES:
Delirium severity within 5 days | Up to 5 days after enrollment
  Delirium severity will be assessed twice daily (8:00-10:00 am, 18:00-20:00 pm) with the Confusion Assessment Method-Severity (CAM-S).
Time to first delirium resolution | Up to 5 days after enrollment
  Delirium resolution indicates no delirium episode for at least 24 hours.
Delirium subtype | Up to 5 days after enrollment
  Each time before assessing delirium, sedation or agitation will be assessed using the Richmond Agitation Sedation Scale (RASS), with scores ranging from -5 (unarousable) to +4 (combative) and 0 indicates alert and calm. Patients with delirium will be classified into three subtypes: hyperactive (RASS consistently positive, from +1 to +4), hypoactive (RASS consistently neutral or negative, from -3 to 0), and mixed.
Length of hospital stay after surgery | Up to 30 days after surgery
  Length of hospital stay after surgery
Quality of life at 30 days after surgery | At 30 days after surgery
  Quality of life will be assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF) which is a 24-item questionnaire that assesses the quality of life in physical, psychological, and social relationship, and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.

OTHER OUTCOMES:
Pain intensity | Up to 5 days after enrollment
  Pain intensity, both at rest and with movement, will be assessed twice daily (8:00-10:00 am, 18:00-20:00 pm) with the numeric rating scale (NRS), an 11-point scale where 0 indicates no pain and 10 the worst pain.
Subjective sleep quality | Up to 5 days after enrollment
  Subjective sleep quality will be assessed once daily (8:00-10:00 am) with the numeric rating scale (NRS), an 11-point scale where 0 indicates the best possible sleep and 10 the worst possible sleep.
Non-delirium complications | Up to 30 days after surgery
  Defined as new-onset medical conditions other than delirium that were deemed harmful and required therapeutic intervention, i.e., grade II or higher on the Clavien-Dindo classification.
All-cause mortality | Up to 30 days after surgery
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital

REFERENCES:
- [Background] Silva AR, Regueira P, Albuquerque E, Baldeiras I, Cardoso AL, Santana I, Cerejeira J. Estimates of Geriatric Delirium Frequency in Noncardiac Surgeries and Its Evaluation Across the Years: A Systematic Review and Meta-analysis. J Am Med Dir Assoc. 2021 Mar;22(3):613-620.e9. doi: 10.1016/j.jamda.2020.08.017. Epub 2020 Oct 1. PMID 33011097
- [Background] Berian JR, Zhou L, Russell MM, Hornor MA, Cohen ME, Finlayson E, Ko CY, Rosenthal RA, Robinson TN. Postoperative Delirium as a Target for Surgical Quality Improvement. Ann Surg. 2018 Jul;268(1):93-99. doi: 10.1097/SLA.0000000000002436. PMID 28742701
- [Background] Rong X, Ding ZC, Yu HD, Yao SY, Zhou ZK. Risk factors of postoperative delirium in the knee and hip replacement patients: a systematic review and meta-analysis. J Orthop Surg Res. 2021 Jan 22;16(1):76. doi: 10.1186/s13018-020-02127-1. PMID 33482875
- [Background] Zhou Q, Zhou X, Zhang Y, Hou M, Tian X, Yang H, He F, Chen X, Liu T. Predictors of postoperative delirium in elderly patients following total hip and knee arthroplasty: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2021 Nov 12;22(1):945. doi: 10.1186/s12891-021-04825-1. PMID 34772392
- [Background] Kitsis P, Zisimou T, Gkiatas I, Kostas-Agnantis I, Gelalis I, Korompilias A, Pakos E. Postoperative Delirium and Postoperative Cognitive Dysfunction in Patients with Elective Hip or Knee Arthroplasty: A Narrative Review of the Literature. Life (Basel). 2022 Feb 20;12(2):314. doi: 10.3390/life12020314. PMID 35207601
- [Background] Lat I, McMillian W, Taylor S, Janzen JM, Papadopoulos S, Korth L, Ehtisham A, Nold J, Agarwal S, Azocar R, Burke P. The impact of delirium on clinical outcomes in mechanically ventilated surgical and trauma patients. Crit Care Med. 2009 Jun;37(6):1898-905. doi: 10.1097/CCM.0b013e31819ffe38. PMID 19384221
- [Background] Quinlan N, Rudolph JL. Postoperative delirium and functional decline after noncardiac surgery. J Am Geriatr Soc. 2011 Nov;59 Suppl 2:S301-4. doi: 10.1111/j.1532-5415.2011.03679.x. PMID 22091577
- [Background] Lescot T, Karvellas CJ, Chaudhury P, Tchervenkov J, Paraskevas S, Barkun J, Metrakos P, Goldberg P, Magder S. Postoperative delirium in the intensive care unit predicts worse outcomes in liver transplant recipients. Can J Gastroenterol. 2013 Apr;27(4):207-12. doi: 10.1155/2013/289185. PMID 23616958
- [Background] Abelha FJ, Luis C, Veiga D, Parente D, Fernandes V, Santos P, Botelho M, Santos A, Santos C. Outcome and quality of life in patients with postoperative delirium during an ICU stay following major surgery. Crit Care. 2013 Oct 29;17(5):R257. doi: 10.1186/cc13084. PMID 24168808
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Swarbrick CJ, Partridge JSL. Evidence-based strategies to reduce the incidence of postoperative delirium: a narrative review. Anaesthesia. 2022 Jan;77 Suppl 1:92-101. doi: 10.1111/anae.15607. PMID 35001376
- [Background] Inouye SK, Bogardus ST Jr, Baker DI, Leo-Summers L, Cooney LM Jr. The Hospital Elder Life Program: a model of care to prevent cognitive and functional decline in older hospitalized patients. Hospital Elder Life Program. J Am Geriatr Soc. 2000 Dec;48(12):1697-706. doi: 10.1111/j.1532-5415.2000.tb03885.x. PMID 11129764
- [Background] Hshieh TT, Yang T, Gartaganis SL, Yue J, Inouye SK. Hospital Elder Life Program: Systematic Review and Meta-analysis of Effectiveness. Am J Geriatr Psychiatry. 2018 Oct;26(10):1015-1033. doi: 10.1016/j.jagp.2018.06.007. Epub 2018 Jun 26. PMID 30076080
- [Background] Morandi A, Brummel NE, Ely EW. Sedation, delirium and mechanical ventilation: the 'ABCDE' approach. Curr Opin Crit Care. 2011 Feb;17(1):43-9. doi: 10.1097/MCC.0b013e3283427243. PMID 21169829
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Sternberg SA, Chandran A, Sikka M. Alternative therapy use by elderly African Americans attending a community clinic. J Am Geriatr Soc. 2003 Dec;51(12):1768-72. doi: 10.1046/j.1532-5415.2003.51562.x. PMID 14687356
- [Background] Ryder PT, Wolpert B, Orwig D, Carter-Pokras O, Black SA. Complementary and alternative medicine use among older urban African Americans: individual and neighborhood associations. J Natl Med Assoc. 2008 Oct;100(10):1186-92. doi: 10.1016/s0027-9684(15)31475-9. PMID 18942280
- [Background] Loera JA, Reyes-Ortiz C, Kuo YF. Predictors of complementary and alternative medicine use among older Mexican Americans. Complement Ther Clin Pract. 2007 Nov;13(4):224-31. doi: 10.1016/j.ctcp.2007.03.002. Epub 2007 Apr 18. PMID 17950177
- [Background] Levy I, Gavrieli S, Hefer T, Attias S, Schiff A, Oliven R, Wisberg-Levi S, Hanchinsky R, Schiff E. Acupuncture Treatment of Delirium in Older Adults Hospitalized in Internal Medicine Departments: An Open-Label Pragmatic Randomized-Controlled Trial. J Geriatr Psychiatry Neurol. 2022 May;35(3):333-343. doi: 10.1177/0891988721996804. Epub 2021 Mar 9. PMID 33685268